CLINICAL TRIAL: NCT01806909
Title: Phase 1 Study of Safety and Immunogenicity of Intranasal Ad4-H5-VTN in Ad4 Seronegative and Seropositive Volunteers
Brief Title: Intranasal AD4-H5-VTN as an Adenovirus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130081; 13-I-0081
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-04-22

CONDITIONS: Healthy Volunteer
Keywords: Flu Vaccine; Healthy Volunteer
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intranasal (Other): Ad4-H5-VTN intranasal vaccine administered in cohorts of 3 at increasing dosages
  Interventions: Biological: Ad4-H5-Vtn

INTERVENTIONS:
Biological: Ad4-H5-Vtn

SUMMARY:
Background:

* Adenoviruses are viruses that typically cause symptoms of a cold or eye infection. These viruses are being tested as part of a possible new vaccine. Researchers hope that the adenovirus will help carry the vaccine into the body and cause an immune response. An immune response is the body s release of cells and substances that protect the body from infection. If an adenovirus vaccine can be developed, it might be used as part of a vaccine for malaria or other serious illnesses. Researchers want to test the adenovirus vaccine as a nasal spray in healthy volunteers. The vaccine is called AD4-H5-VTN.
* Because the vaccine contains a live adenovirus, there is a possibility that participants can infect other people. Therefore, participants' intimate contacts must join this study. An intimate contact is someone who the participant will kiss on the mouth or have sexual intercourse with during the period of this study.

Objectives:

* To study the immune response of the AD4-H5-VTN vaccine in healthy volunteers.
* To see if the adenovirus in the AD4-H5-VTN vaccine is contagious or spreads to others.

Eligibility:

* Healthy volunteers between 18 and 49 years of age.
* Intimate contacts of healthy volunteers between 18 and 65 years of age.
* Participants must not have evidence of previous exposure to adenovirus type 4.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants who will receive the vaccine must be willing to be hospitalized for between 5 and 7 days. They will come to the National Institutes of Health for follow-up visits weekly for the first month, after 8 weeks, in 6 months, and possibly 1 year. They must also avoid all vaccines (including seasonal flu vaccine) and allergy shots for 30 days before and after having the study vaccine.
* Participants will enter the hospital for the vaccine study visit. They will receive the vaccine as a nasal spray. Because the vaccine uses a live virus, participants may be contagious for the virus for up to 4 weeks. They will remain in the hospital in respiratory isolation for 7 days, or until they have two negative nasal washes taken 1 day apart. A negative nasal wash means that there is no live virus in the nose.
* After leaving the hospital, participants will keep a diary at home for at least 3 weeks. They will record their temperature, any symptoms, or other health changes every day during this time.
* Participants should avoid intimate contact with others for 28 days after having the vaccine. Intimate contact includes kissing on the mouth and sexual intercourse. Also, participants should not share kitchen utensils, drinking cups, towels, or hair combs with others. Intimate contacts will also keep track of any illnesses or symptoms they develop during this time.
* At the follow-up visits, participants will provide blood and swab samples for study.

DETAILED DESCRIPTION:
This is a Phase 1 single center, dose-escalation study designed to evaluate the safety and immunogenicity of live, replication competent recombinant Adenovirus type 4-H5N1 Influenza Vietnam 1194 Hemagglutinin (HA) (Ad4-H5-Vtn). Determining the optimal route and dose for this recombinant platform will greatly accelerate investigations of this vector as an influenza vaccine and an HIV vaccine platform.

The primary goal of this study is to evaluate safety of ascending dosages of the Ad4-H5-Vtn vaccine following intranasal administration. A dosage will be selected to further evaluate the humoral, cellular, and mucosal immune responses against both the vector and the inserted gene. The Ad4-H5-Vtn will be initiated at 103 viral particles (vp). Once safety is established at the initial dose, a second round of testing will begin at the next ten-fold higher dose. The Ad4-H5-Vtn vaccine will be assessed in three participants at each dosage level. The maximum viral dose administered will be 108 vp.

In addition to clinical and laboratory monitoring of safety, the principal assessments will be shedding of the Ad4-H5-Vtn virus in rectal, cervicovaginal, throat, and nasal swabs, and assessment of the antibody (mucosal and systemic) response to the HA and to the Ad4 virus. Participants will remain in the NIH Special Clinical Studies Unit until they have 2 consecutive negative nasal washes or 7 days have elapsed since vaccination, whichever occurs first; they may remain on the unit longer if medically necessary. When safety has been confirmed in all 3 participants at a given dosage level, the next higher dose group is enrolled. If one grade 3 or greater toxicity (or pre-specified grade 2 toxicity, see Section 3.4) at least possibly related to the vaccine is observed, the group will be expanded at that dose. If a second at least possibly related grade 3 or greater toxicity (or pre-specified Grade 2 toxicity, see Section 3.4) is observed, the dose will be reduced one level and the group will be expanded. Up to 25 Ad4-seronegative individuals will be enrolled at the maximum tolerated dose to fully evaluate safety and immunogenicity in the protocol.

All participants will be followed for 28 days following immunization, and again at 8 and 26 weeks to evaluate any long-term toxicity and persistence of immunity. All subjects will be offered to receive a booster vaccine at the 26-week visit and be seen for follow-up visits 4 and 8 weeks following booster immunization with an additional telephone follow-up 6 months after boosting. Household and intimate contacts will also be enrolled and monitored for Adenovirus and HAI antibodies following Ad4-H5-Vtn administration only; household and intimate contacts will not be enrolled or monitored during the boost portion of the study.

We will conduct an expansion H5N1 boost phase of this study, in which all vaccinees from the initial phase of the study will be offered re-enrollment to receive a booster vaccination with an FDA-approved H5N1 inactivated monovalent influenza vaccine. We will offer enrollment in the expansion phase to all participants who received the Ad4-H5-Vtn vaccine in the initial phase, regardless of whether they also received the recombinant hemagglutinin influenza H5 vaccine boost. We will also enroll individuals who have never received an H5 influenza vaccine as controls. Participants will receive a single vaccination with the H5N1 vaccine and be seen for follow-up visits 4 and 8 weeks later for immunogenicity evaluations.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participant (vaccinees, household contacts, and intimate contacts) must meet all of the following criteria:

1. Age 18 to 49 years for vaccinees. Vaccinnees may be greater than 49 years of age at the time of booster vaccination. Age 18 to 65 years for household and intimate contacts.
2. Able to provide proof of identity to the acceptance of the Principal Investigator or designee during enrollment.
3. Available and willing to participate in follow-up visits and tests for the duration of the study.
4. Willing to have samples stored for future research

The following inclusion criteria apply to vaccines and intimate contacts, but not to household contacts:

1. In good general health without clinically significant medical history.
2. Negative b-HCG pregnancy test for females presumed to be of reproductive potential.
3. A female must meet one of the following criteria:

   1. No reproductive potential because of menopause (one year without menses) or because of a hysterectomy, bilateral oophorectomy, or tubal ligation.
   2. Participant agrees to be heterosexually inactive or consistently practice contraception at least 21 days prior to enrollment and 28 days following vaccination. Acceptable methods of contraception include the following:

      * condoms, male or female, with a spermicide
      * diaphragm or cervical cap with spermicide
      * contraceptive pills, Norplant, or Depo-Provera
      * male partner has previously undergone a vasectomy for which there is documentation.
      * intrauterine device
4. Male participants must agree to practice abstinence or effective birth control for at least 21 days prior to enrollment and during the first 28 days following vaccination.

The following inclusion criteria apply only to vaccinees and not to household or intimate contacts:

1. Willing to receive HIV test results and abide by NIH guidelines for partner notification of positive HIV results.
2. Physical examination and laboratory results without clinically significant findings within the 8 weeks prior to enrollment.
3. Willing to avoid vaccination other than the study agent for 30 days prior to and 30 days after administration of the Ad4-H5-Vtn vaccine.
4. Safety Laboratory Criteria within 8 weeks prior to enrollment:

   Hematopoietic: White blood cell count and Lymphocyte count +/- 25% the normallimits for the NIH Clinical Center
   * Platelet count of least 125,000/mm(3)
   * Hemoglobin greater than 11.2 g/dL for females and greater than 13.0 g/dL for males.
   * Renal: BUN less than 23 mg/dL; creatinine within normal limits for the NIH Clinical Center
   * Hepatic: Serum total bilirubin less than or equal to 2 mg/dL
   * Metabolic: ALT < 2 times upper limit of normal range
   * Endocrine: Serum glucose within normal range
5. Additional Laboratory Criteria:

   * Immunologic: No history of hypogammaglobulinemia
   * Serologic: Ad4 neutralizing antibody 80% inhibitory dilution less than 1:100 ((This criterion does not apply to participants in vaccine arm B.)
6. Willing to be hospitalized at the Clinical Center under respiratory precautions for up to 7 days or longer if medically indicated.

Inclusion criteria for the expansion H5N1 boost phase:

1. Age 18 to 64.
2. Negative pregnancy test (women of childbearing potential).
3. Group-specific inclusion criteria:

   * For participants in the study group: prior receipt of the Ad4-H5-Vtn vaccine in the initial phase of this study.
   * For participants in the control group: no prior receipt of an H5 vaccine product (by self-report).

EXCLUSION CRITERIA:

A participant (vaccinees, household contacts, and intimate contacts) will be excluded if they have the following:

1. Any condition that, in the investigator s judgement, places the subject at undue risk by participating in the study.

The following exclusion criterion applies to vaccines and intimate contact, but not to household contacts:

1. History of any prior disease or therapy which would affect immune or pulmonary function.
2. Prior malignancy, except curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
3. History of radiation therapy or cytotoxic/cancer chemotherapy.
4. History of diabetes mellitus.
5. Immunodeficiency or autoimmune disease.
6. Acute infection or a recent (within 6 months) history of chronic infection suggestive of immunodeficiency.
7. Taking any medication which may affect immune function, except participants may be taking low doses of nonprescription strength NSAIDS (including e.g. ibuprofen or aspirin) or acetaminophen.
8. Chronic respiratory disorders including asthma, emphysema, interstitial lung disease, pulmonary hypertension, recurrent pneumonia, or recent or ongoing respiratory tract infection. If a respiratory disorder is transient, defer immunization but do not exclude the participant.
9. Active Hepatitis B or C infection (i.e. Hepatitis B or C positive serology with the presence of virus antigen or DNA. Ongoing viral replication will be confirmed by a Hepatitis B antigen or Hepatitis C viral load).
10. Female of child-bearing potential who is breast-feeding or planning pregnancy during the 28 days following vaccination.

The following exclusion criteria apply only to vaccinees and not to household or intimate contacts:

1. Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to receipt of live virus vaccine, protocol adherence, or a participant s ability to give informed consent.
2. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to

   enrollment.
3. Participants that live in the same house or apartment with any of the following will be excluded:

   1. An individual under 18 years of age
   2. An immunocompromised or immunosuppressed individual
   3. An individual with chronic respiratory disease
   4. A woman who is currently pregnant or planning a pregnancy during the period of immunization
4. Healthcare worker who has direct contact with immunodeficient, unstable patients, or pediatric patients.
5. Participants caring for children less than 36 months of age.
6. Receipt of any of the following:

   * Antiviral medications within 30 days prior to vaccination
   * Blood products within 120 days prior to HIV screening
   * Immunoglobulin within 60 days prior to HIV screening
   * Investigational research drugs or any other investigational agent that in the judgement of the PI might interact with the study vaccine within 30 days prior to initial study vaccine administration
   * Allergy treatment with antigen injections within 30 days of study vaccine administration
7. History of Guillain-Barr(SqrRoot)(Copyright) syndrome.
8. History of H5 influenza vaccination. (This criterion does not apply to participants in vaccine arm B.)

Exclusion criteria for the expansion H5N1 boost phase:

1. History of systemic hypersensitivity reactions to egg proteins or life-threatening reactions to previous influenza vaccinations.
2. History of Guillain-Barr(SqrRoot)(Copyright) syndrome.
3. Acute infection or a recent (within 6 months) history of chronic infection suggestive of immunodeficiency.
4. Taking any medication which may affect immune function, except participants may be taking low doses of nonprescription strength NSAIDS (including e.g. ibuprofen or aspirin) or acetaminophen.
5. Receipt of an approved vaccine, investigational research drugs, or any other investigational agent that in the judgement of the PI might interact with the study vaccine within 30 days prior to H5N1 vaccine administration.
6. Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to receipt of the H5N1 vaccine, protocol adherence, or a participant s ability to give informed consent.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-03-06; Primary Completion 2018-01-09 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the Ad4-H5-Vtn recombinant vaccine in Ad4 seronegative humans when administered intranasally | Ongoing

SECONDARY OUTCOMES:
To evaluate the immunogenicity of the Ad4-H5-Vtn recombinant vaccine in Ad4 seronegative humans when administered intranasally | Months 2, 6
To determine the optimal dose for the nasal Ad4 vaccine platform, up to a maximum dose of 108 vp. | Ongoing
To monitor transmission to household and intimate contacts of vaccines and To monitor shedding and stability of recovered Ad4 recombinants. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Mark Connors, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Connors M, Collins PL, Firestone CY, Sotnikov AV, Waitze A, Davis AR, Hung PP, Chanock RM, Murphy BR. Cotton rats previously immunized with a chimeric RSV FG glycoprotein develop enhanced pulmonary pathology when infected with RSV, a phenomenon not encountered following immunization with vaccinia--RSV recombinants or RSV. Vaccine. 1992;10(7):475-84. doi: 10.1016/0264-410x(92)90397-3. PMID 1609551
- [Background] Couch RB, Cate TR, Fleet WF, Gerone PJ, Knight V. Aerosol-induced adenoviral illness resembling the naturally occurring illness in military recruits. Am Rev Respir Dis. 1966 Apr;93(4):529-35. doi: 10.1164/arrd.1966.93.4.529. No abstract available. PMID 4286394
- [Background] Edmondson WP, Purcell RH, Gundelfinger BF, Love JW, Ludwig W, Chanock RM. Immunization by selective infection with type 4 adenovirus grown in human diploid tissue culture. II. specific protective effect against epidemic disease. JAMA. 1966 Feb 7;195(6):453-9. No abstract available. PMID 4285433
- [Derived] Matsuda K, Migueles SA, Huang J, Bolkhovitinov L, Stuccio S, Griesman T, Pullano AA, Kang BH, Ishida E, Zimmerman M, Kashyap N, Martins KM, Stadlbauer D, Pederson J, Patamawenu A, Wright N, Shofner T, Evans S, Liang CJ, Candia J, Biancotto A, Fantoni G, Poole A, Smith J, Alexander J, Gurwith M, Krammer F, Connors M. A replication-competent adenovirus-vectored influenza vaccine induces durable systemic and mucosal immunity. J Clin Invest. 2021 Mar 1;131(5):e140794. doi: 10.1172/JCI140794. PMID 33529172